CLINICAL TRIAL: NCT00755768
Title: More Time Better Outcome - a Randomised Trial to Investigate the Effect of More Dietetic Time on Phosphate Levels in End Stage Renal Failure Patients
Brief Title: More Time Better Outcome - a Randomised Trial to Investigate the Effect of More Dietetic Time in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Free Hampstead NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 05/Q0504/46; BRS grant; R&D 7119M; NCT00454727 (obsolete NCT alias)
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Renal Failure
Keywords: hemodialysis; phosphate; calcium phosphate product; dietician; dietetic advice
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: additional review by dietician

SUMMARY:
The purpose of this study is to determine whether spending more time with a dietitian will improve dietary compliance in a group of hemodialysis patients, with particular respect to phosphate control.

DETAILED DESCRIPTION:
* randomised prospective controlled trial
* stable haemodialysis patients on thrice weekly haemodialysis (URR > 66%)
* either had standard dietetic review - 6 monthly or intensive review - monthly
* all patients had to have a serum phosphate > 1.8 mmol/l over the previous three months to be recruited
* study period 6 months, and then patients followed for a further 3 months

ELIGIBILITY:
Inclusion Criteria:

* stable chronic hemodialysis patients
* serum phosphate > 1.8 mmol/l sustained over 3 months prior to trial entry adequate dialysis treatment as assessed by urea reduction

Exclusion Criteria:

* pregnancy
* unable to give consent
* phosphate < 1.8 mmol/l
* inadequate dialysis
* aged < 18 or > 80
* poor nutritional state
* weight loss in proceeding three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2006-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
phosphate control
calcium phosphate product

SECONDARY OUTCOMES:
parathyroid hormone
number and type of phosphate binders prescribed

CONTACTS AND LOCATIONS:
Overall Officials: andrew davenport, md, Principal Investigator — UCL Center for nephrology
Locations (1):
- UCL Center for Nephrology, London, London, United Kingdom